CLINICAL TRIAL: NCT04451967
Title: the Acute Myocardial Infarction Study in Northeastern China
Brief Title: Acute Myocardial Infarction Study in Northeastern China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Hospital of Jilin University (Other)
Collaborators: Yanbian University Hospital (Unknown); Dunhua City Hospital in Jilin Province (Unknown); Liaoyuan City Central Hospital (Unknown); Dongliao People's Hospital (Unknown); Songyuan Central Hospital (Unknown); Changling People's Hospital (Unknown); Siping Central People's Hospital (Other); The First People's Hospital of Manchu Autonomous County (Unknown); Changchun Center Hospital (Unknown); Nongan People's Hospital (Unknown); Beihua University (Other); Jilin Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Panshi City Hospital (Unknown); Tonghua Central Hospital (Unknown); Baishan Central Hospital (Unknown); Jingyu People's Hospital (Unknown); Meihekou Central Hospital (Unknown); Baicheng Central Hospital (Unknown); Tongyu First Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: SecondJilinU-AMINoC
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transfer after thrombolysis
  Interventions: Procedure: thrombolysis
- Transfer after DAPT
- Direct transfer

INTERVENTIONS:
Procedure: thrombolysis — transfer after thrombolysis for STEMI patients within 6h since onset
  Other Names: DAPT
  Groups: Transfer after thrombolysis

SUMMARY:
This is a real-world prospective cohort study aiming to generate knowledge about the characteristics, treatments, and outcomes of hospitalized AMI patients in Jilin Province. The study includes hospitalizations diagnosed of AMI, including ST segment-elevation myocardial infarction (STEMI) and non-ST-segment-elevation myocardial infarction (NSTEMI).

ELIGIBILITY:
Inclusion Criteria:

* patients admitted within 7 days of acute myocardial ischemic symptoms with a primary clinical diagnosis of AMI, meet Fourth Universal Definition for Myocardial Infarction (2018)

Exclusion Criteria:

* Types 4a and type 5 AMI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients must be admitted within 7 days of acute myocardial ischemic symptoms with a primary clinical diagnosis of AMI, including ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI). Final inclusion criteria must meet Fourth Universal Definition for Myocardial Infarction (2018)
Sampling Method: Probability Sample
Enrollment: 3159 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-09-09 (Estimated); Study Completion 2022-09-09 (Estimated)

PRIMARY OUTCOMES:
all-cause death | 2 years post discharge
  all-cause death

SECONDARY OUTCOMES:
major adverse cardiac events (MACE) | 2 years post discharge
  recurrent angina, non-fatal myocardial infarction, cardiac failure, malignant arrhythmia, and death from cardiovascular causes

CONTACTS AND LOCATIONS:
Overall Officials: Bin Liu, Ph.D, Principal Investigator — Second Hospital of Jilin University
Locations (1):
- The second hospital of Jilin university, Changchun, Jilin, China

REFERENCES:
- [Derived] Li T, Wu J, Liu J, Sun W, Qi C, Liu B, Wells GA, Wang J; Acute Myocardial Infarction Study in Northeastern China (AMINoC). Protocol for the Acute Myocardial Infarction Study in Northeastern China (AMINoC): a real-world prospective cohort study. BMJ Open. 2021 May 25;11(5):e042936. doi: 10.1136/bmjopen-2020-042936. PMID 34035090